CLINICAL TRIAL: NCT07142421
Title: A Phase II Clinical Study of Trifluridine/Tipiracil Combined With Anlotinib as Second-line Treatment for Recurrent and Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: A Study of Trifluridine/Tipiracil Combined With Anlotinib as Second-line Treatment for Recurrent and Metastatic Esophageal Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, QiangfengWang, Principal Investigator, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2025C]IIT. No.123
Record Dates: First submitted 2025-08-10; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: escc; second-line treatment; Anlotinib; Trifluridine and Tipiracil
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Combined Modality Therapy; trifluridine tipiracil drug combination; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trifluridine/tipiracil combined with Anlotinib Group (Experimental): Trifluridine/tipiracil combined with Anlotinib for second-line treatment of recurrent and metastatic ESCC
  Interventions: Drug: Combination therapy (COMB)

INTERVENTIONS:
Drug: Combination therapy (COMB) — Trifluridine/tipiracil combined with Anlotinib in treatment
  Other Names: Trifluridine/tipiracil; Anlotinib

SUMMARY:
Esophageal squamous cell carcinoma (ESCC) is one of the malignant tumors with a high incidence worldwide, especially remaining persistently high in Asian regions. Despite advancements in early diagnosis and comprehensive treatment, most patients are already in the locally advanced or metastatic stage at the time of initial diagnosis, resulting in an extremely poor prognosis. The objective response rate (ORR) of first-line chemotherapy regimens (such as platinum-containing dual-drug combinations with fluorouracil) is less than 50%, and the median progression-free survival (PFS) is only 3-6 months. Moreover, the options for second-line treatment are more limited. Currently, there is no unified standard for second-line treatment, and there is an urgent need to explore new and effective regimens.

Anlotinib is a multi-target tyrosine kinase inhibitor that can target and inhibit vascular endothelial growth factor receptor (VEGFR), fibroblast growth factor receptor (FGFR), and platelet-derived growth factor receptor (PDGFR). It exerts anti-tumor effects through anti-angiogenesis and regulation of the tumor microenvironment. Single-agent anlotinib has shown certain efficacy in advanced esophageal cancer. A phase II study indicated that the ORR of single-agent anlotinib in second-line treatment was 9.7%, with a median PFS of 3.0 months.

Suyuan (trifluridine/tipiracil) is a new oral fluoropyrimidine drug composed of trifluridine (a cytotoxic component) and tipiracil (a synergist that inhibits the metabolic enzyme TP), which can overcome the resistance to traditional fluorouracil. Single-agent Suyuan has achieved significant survival benefits in metastatic colorectal cancer, and its synergistic effect in combination with anti-angiogenic drugs in solid tumors has also been preliminarily confirmed.

The biological basis of combination therapy: Anti-angiogenic drugs can improve the hypoxic state of the tumor microenvironment, enhance the delivery efficiency of chemotherapy drugs, and simultaneously inhibit the infiltration of immunosuppressive cells. Their combination with chemotherapy or immunotherapy has potential synergistic effects. Preclinical studies have shown that anlotinib combined with fluoropyrimidine drugs can significantly inhibit the growth of esophageal cancer models by dual inhibition of tumor proliferation and angiogenesis pathways.

Based on the above background, this study intends to explore the efficacy and safety of Suyuan combined with anlotinib in the second-line treatment of recurrent and metastatic ESCC, aiming to provide new treatment options for patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed esophageal squamous cell carcinoma.
2. Clinical stage IIIB-C or IV according to the 8th edition of AJCC.
3. Having at least one measurable or evaluable lesion.
4. ECOG performance status score of 0-2.
5. Failed first-line standard treatment regimens.
6. Age ≥ 18 years.
7. Normal function of major organs.
8. Female subjects of childbearing age must undergo a pregnancy test within 3 days before the first dose with a negative result, and adopt effective contraceptive measures during the study period.

Exclusion Criteria:

1. Patients with other malignant tumors requiring treatment.
2. Patients with severe diseases of major organs such as heart, liver, and kidney.
3. Patients who have previously received treatment with anti-angiogenic monoclonal antibodies or small-molecule tyrosine kinase inhibitors.
4. Patients with an expected survival period of < 3 months.
5. Patients who have previously used fluoropyrimidine drugs (such as 5-FU, capecitabine, etc.).
6. Patients with Uncontrolled active infections (such as HIV, HCV, HBV, etc.).
7. Pregnant or lactating women.
8. Other circumstances deemed unsuitable for enrollment by the researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From date of therapy until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The time interval from the day a patient starts receiving a certain treatment (or is randomized into a treatment regimen) to the occurrence of objective tumor progression (or death from any cause).

SECONDARY OUTCOMES:
Overall Survival (OS) | From date of therapy until the date of death, assessed up to 24 months
  OS focuses on the time from the start of treatment to the patient's death (regardless of the cause)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No